CLINICAL TRIAL: NCT01544322
Title: Phase 1 Open Label Dose Escalation Study of the Safety and Pharmacokinetics of ME-344 as a Single Agent in Patients With Refractory Solid Tumors
Brief Title: Dose Escalation Study of the Safety and Pharmacokinetics of ME-344 Single Agent for Refractory Solid Tumors
Acronym: ME-344-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MEI Pharma, Inc. (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-344-001
Record Dates: First submitted 2012-02-22; First posted 2012-03-05 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2014-04

CONDITIONS: Solid Tumors
Keywords: solid tumors; recurrent; advanced; metastatic; refractory
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — ME-344; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ME-344 — experimental drug, dose escalation with 5 planned dose cohorts of 1.2 mg/kg, 2.5 mg/kg, 5 mg/kg, 10 mg/kg, 20 mg/kg; Cycle 1 is 3 weekly IV infusions on Days 1, 8, and 15. After safety assessment, if there is clinical benefit, weekly dosing may continue until withdrawal.
  Once the highest tolerated dose has been determined, patients will be enrolled to receive IV infusions 2 days each week. Cycle 1 at the highest dose level is 3 weekly IV infusions on days 1, 2, 8, 9, 15 and 16. After safety assessment, if there is clinical benefit, weekly dosing may continue until withdrawal.
  Other Names: open label; single agent

SUMMARY:
The purpose of this study is to determine the tolerability of ME-344, find the maximum tolerated dose, and the safety profile in patients with refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Male or female ≥ 18 years of age
* Histologic or cytologic confirmed locally advanced or metastatic cancer that has no standard therapeutic alternatives.
* ECOG Performance status 0-1 (Appendix A)
* A minimum life expectancy of 12 weeks
* Adequate bone marrow, hepatic and renal function as evidenced by:

  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * Platelet count > 100 x 109/L
  * Hemoglobin > 9.0 g/dL
  * Serum bilirubin < 1.5 x ULN
  * AST/ALT (SGOT/SGPT) < 2.5 x ULN for the reference laboratory or < 5 x ULN in the presence of liver metastases
  * Serum creatinine < 1.5 x ULN
* Adequate cardiac function as evidenced by:

  * CK-MB within normal levels at baseline
  * Troponin T within normal levels at baseline
  * The average QTc from triplicate screening ECGs (every 5 minutes over a total of 15 minutes) must be < 470 msec to be eligible for the study. (If a patient has an average QTc interval >470 msec at screening, the screening ECG may be repeated twice (at least 24 hours apart).
  * LV Ejection Fraction > lower limit of institutional normal level
* All potentially fertile patients will agree to use an effective form of contraception during the study and for 30 days following the last dose of ME-344 (an effective form of contraception is defined as an oral contraceptive or a double barrier method).
* At least 4 weeks must have elapsed prior to Day 1 Cycle 1 since prior chemotherapy (6 weeks for nitrosourea or mitomycin C), investigational drug or biologic therapy and any toxicity associated with these treatments has recovered to ≤ NCI-CTCAE Grade 1.
* At least 21 days must have elapsed prior to Day 1 Cycle 1, radiotherapy, immunotherapy or following major surgery and any surgical incision should be completely healed. At least 14 days must have elapsed prior to Day 1 Cycle 1 for "limited palliative radiotherapy", defined as a course of therapy encompassing <25% total bone marrow volume and not exceeding 30 Gy.

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Tumor involvement of the Central Nervous System (CNS):

  * Patients with treated and stable CNS metastases may be eligible to participate after discussion and approval from the Medical Monitor
* Uncontrolled infection or systemic disease.
* Clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease e.g. angina, and cardiac arrhythmias) or myocardial infarction within the last 12 months.
* Any major surgery, radiotherapy, or immunotherapy within the last 21 days. Limited palliative radiation, defined as encompassing <25% of total bone marrow volume and not exceeding a total dose of 30 Gy, within the last 14 days.
* Chemotherapy regimens with delayed toxicity within the last 4 weeks (or within 6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential or delayed toxicity within the last 2 weeks.
* No concurrent systemic chemotherapy or biologic therapy is allowed.
* Known hypersensitivity to any components of ME-344 study drug product.
* Known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both).
* History of solid organ transplantation.
* Psychiatric disorder or social or geographic situation that would preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | One Cycle of 28 days
  Patients will be administered ME-344 IV infusions weekly for 3 weeks during the first 28 days cycle for dose limiting toxicity. Patients will be assessed by physical exam, vital signs, hematology and clinical chemistry, urinalysis, ECG, echocardiogram and pharmacokinetic sampling.

SECONDARY OUTCOMES:
Response Rate | baseline and a minimum of every 12 weeks
  Radiologic assessments will be performed at baseline and a minimum of every 12 weeks. Patients may continue weekly dosing if there is clinical beneficial determined by the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Mass, MD, Study Chair — MEI Pharma, Inc.
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- See also: Sponsor's web site — http://marshalledwardsinc.com